CLINICAL TRIAL: NCT02518672
Title: Role of DHA Monoglyceride (MAG-DHA) in the Resolution of Pulmonary Inflammation of Patients With Cystic Fibrosis.
Brief Title: Pro-resolving Effect of MAG-DHA in Cystic Fibrosis (PREMDIC)
Acronym: PREMDIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SCF Pharma (Industry)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Solutex GC S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-108
Record Dates: First submitted 2015-08-03; First posted 2015-08-10 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — docosahexaenoic acid monoacylglyceride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAG-DHA (Active Comparator): MAG-DHA 8 x 625 mg softgels by mouth, every day at bedtime for 90 days.
  Interventions: Dietary Supplement: MAG-DHA
- Placebo (Placebo Comparator): Placebo (sunflower oil) 8 x 625 mg softgels by mouth, every day at bedtime for 90 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MAG-DHA — MAG-DHA 8 x 625 mg softgels by mouth, every day at bedtime for 90 days.
  Arms: MAG-DHA
Dietary Supplement: Placebo — Placebo (sunflower oil) 8 x 625 mg softgels by mouth, every day at bedtime for 90 days.
  Arms: Placebo

SUMMARY:
Monoglyceride of DHA (DHA-MAG) is a lipid compound for which intestinal absorption would increase the ratio DHA / arachidonic acid (AA) and promote the synthesis of specific metabolites involved in the resolution of inflammation.

The PREMDIC project, initiated at the Centre Hospitalier Universitaire de Sherbrooke, is a randomized double-blind study for people with cystic fibrosis (CF) and aims to evaluate whether daily supplementation monoglyceride of DHA (a fatty acid omega-3 family) will reduce lung inflammation and improve pulmonary function.

DETAILED DESCRIPTION:
The goal of the study is:

To investigate the efficacity of oral administration of MAG-DHA to increase DHA bioavailability and reduce lung inflammation of patients with cystic fibrosis

The specific objectives of the project are :

* Determine the effect of MAG-DHA on lipid membranes of the blood mononuclear cells.
* Evaluate the effect of MAG-DHA on lung inflammation (determination of Human leukocyte elastase and alpha1 antitrypsin complexes : pHLE).

For this study, 20 cystic fibrosis patients are recruited. Patients are divided into 2 groups of 10 and received a daily dose equivalent to 3 g of placebo (sunflower oil) or MAG-DHA.

The project takes place over a period of 3 months and patients must travel to the research center for a total of five visits including recruitment.

For the 2 groups, DHA ratio / AA is measured in membranes of mononuclear cells. Forced expiratory volume in 1 second (FEV1) is determined and pHLE complexes are detected in plasma as a marker of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. forced expiratory volume in 1 second (FEV1) between 30 - 90%.
2. no respiratory exacerbations during the last 2 weeks before the start of the study
3. not have clotting problems or a history of bleeding diathesis
4. patients with liver function abnormalities are included in the study

Exclusion Criteria:

1. pregnant women or those not using contraception.
2. known allergy to fish and / or seafood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Lung and systemic inflammation measurement | 0 and 90 days
  Docosahexaenoic acid (DHA) and metabolites lipid analyses in plasma and red blood cells Human leukocyte elastase and alpha1 antitrypsin complexes detection in plasma Pulmonary function test (spirometry): Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC) Leukocytes differential cell counts and C reactive protein (CRP) determination level in blood

SECONDARY OUTCOMES:
follow up of vital signs | 0 and 90 days
  weight (Kg)
follow up of vital signs | 0 and 90 days
  Body Mass Index (BMI, Kg/cm2)
follow up of vital signs | 0 and 90 days
  Blood Pressure (mmHg)
lipid profile | 0 and 90 days
  triglycerides (mmol/l)
lipid profile | 0 and 90 days
  cholesterol (mmol/l)
lipid profile | 0 and 90 days
  high density lipoprotein (mmol/l)
lipid profile | 0 and 90 days
  low density lipoprotein (mmol/l)
hepatic function | 0 and 90 days
  measurement of Alanine aminotransferase (ALT) in plasma (U/l)
hepatic function | 0 and 90 days
  measurement of Aspartate aminotransferase (AST) in plasma (U/l)
hepatic function | 0 and 90 days
  measurement of Gamma glutamyl transpeptidase in plasma (U/l)

CONTACTS AND LOCATIONS:
Overall Officials: André M Cantin, M.D., Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Al-Turkmani MR, Freedman SD, Laposata M. Fatty acid alterations and n-3 fatty acid supplementation in cystic fibrosis. Prostaglandins Leukot Essent Fatty Acids. 2007 Nov-Dec;77(5-6):309-18. doi: 10.1016/j.plefa.2007.10.009. Epub 2007 Nov 26. PMID 18036797
- [Background] Andersson C, Al-Turkmani MR, Savaille JE, Alturkmani R, Katrangi W, Cluette-Brown JE, Zaman MM, Laposata M, Freedman SD. Cell culture models demonstrate that CFTR dysfunction leads to defective fatty acid composition and metabolism. J Lipid Res. 2008 Aug;49(8):1692-700. doi: 10.1194/jlr.M700388-JLR200. Epub 2008 Apr 25. PMID 18441018
- [Background] Cantin A. Cystic fibrosis lung inflammation: early, sustained, and severe. Am J Respir Crit Care Med. 1995 Apr;151(4):939-41. doi: 10.1164/ajrccm.151.4.7697269. No abstract available.
- [Background] Dyerberg J, Madsen P, Moller JM, Aardestrup I, Schmidt EB. Bioavailability of marine n-3 fatty acid formulations. Prostaglandins Leukot Essent Fatty Acids. 2010 Sep;83(3):137-41. doi: 10.1016/j.plefa.2010.06.007. PMID 20638827
- [Background] Fortin S, Compositions comprising polyunsaturated fatty acid monoglycerides or derivatives thereof and uses thereof, US819690, 2012, US8222295, 2012.
- [Background] Fortin S, Polyunsaturated fatty acid monoglycerides, derivatives, and uses thereof, CA2672513, 2008, CA2677670, 2010, US8119690, 2011.
- [Background] Freedman SD, Katz MH, Parker EM, Laposata M, Urman MY, Alvarez JG. A membrane lipid imbalance plays a role in the phenotypic expression of cystic fibrosis in cftr(-/-) mice. Proc Natl Acad Sci U S A. 1999 Nov 23;96(24):13995-4000. doi: 10.1073/pnas.96.24.13995. PMID 10570187
- [Background] Mimoun M, Coste TC, Lebacq J, Lebecque P, Wallemacq P, Leal T, Armand M. Increased tissue arachidonic acid and reduced linoleic acid in a mouse model of cystic fibrosis are reversed by supplemental glycerophospholipids enriched in docosahexaenoic acid. J Nutr. 2009 Dec;139(12):2358-64. doi: 10.3945/jn.109.110999. Epub 2009 Oct 14. PMID 19828687
- [Background] Morin C, Fortin S, Cantin AM, Rousseau E. Docosahexaenoic acid derivative prevents inflammation and hyperreactivity in lung: implication of PKC-Potentiated inhibitory protein for heterotrimeric myosin light chain phosphatase of 17 kD in asthma. Am J Respir Cell Mol Biol. 2011 Aug;45(2):366-75. doi: 10.1165/rcmb.2010-0156OC. Epub 2010 Nov 5. PMID 21057106
- [Background] Morin C, Fortin S, Cantin AM, Sirois M, Sirois C, Rizcallah E, Rousseau E. Anti-cancer effects of a new docosahexaenoic acid monoacylglyceride in lung adenocarcinoma. Recent Pat Anticancer Drug Discov. 2013 Sep;8(3):319-34. doi: 10.2174/1574891x113089990032. PMID 23092161
- [Background] Panchaud A, Sauty A, Kernen Y, Decosterd LA, Buclin T, Boulat O, Hug C, Pilet M, Roulet M. Biological effects of a dietary omega-3 polyunsaturated fatty acids supplementation in cystic fibrosis patients: a randomized, crossover placebo-controlled trial. Clin Nutr. 2006 Jun;25(3):418-27. doi: 10.1016/j.clnu.2005.10.011. Epub 2005 Dec 2. PMID 16325968
- [Background] Pier G, Prince A, Cantin A. Cystic fibrosis: an-ion transport issue? Nat Med. 2011 Feb;17(2):166-7. doi: 10.1038/nm0211-166. PMID 21297610
- [Background] Vij N, Mazur S, Zeitlin PL. CFTR is a negative regulator of NFkappaB mediated innate immune response. PLoS One. 2009;4(2):e4664. doi: 10.1371/journal.pone.0004664. Epub 2009 Feb 27. PMID 19247502
- [Result] Cantin AM, Bilodeau G, Larivee P, Richter MV. Plasma biomarkers and cystic fibrosis lung disease. Clin Invest Med. 2012 Jul 4;35(4):E173-81. doi: 10.25011/cim.v35i4.17145. PMID 22863555
- [Result] Morin C, Cantin AM, Rousseau E, Sirois M, Sirois C, Rizcallah E, Fortin S. Proresolving Action of Docosahexaenoic Acid Monoglyceride in Lung Inflammatory Models Related to Cystic Fibrosis. Am J Respir Cell Mol Biol. 2015 Oct;53(4):574-83. doi: 10.1165/rcmb.2014-0223OC. PMID 25781052
- [Derived] Morin C, Cantin AM, Vezina FA, Fortin S. The Efficacy of MAG-DHA for Correcting AA/DHA Imbalance of Cystic Fibrosis Patients. Mar Drugs. 2018 May 26;16(6):184. doi: 10.3390/md16060184. PMID 29861448